CLINICAL TRIAL: NCT07090564
Title: Treatment Outcomes in PASC Patients With Neurocognitive Impairment
Status: Completed | Type: Observational
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Andrew Schamess, MD, Ohio State University
Other Study IDs: 2022H0258
Record Dates: First submitted 2025-07-21; First posted 2025-07-29 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Long COVID
Keywords: Long COVID; PASC; Post-Acute Sequelae of COVID19
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with neurocognitive symptoms receiving care at a Long COVID clinic: OSUMC started a specialized multidisciplinary PASC clinic in March of 2021 to see patients suffering from persistent symptoms after COVID19 infection. The clinic is based in the Division of General Internal Medicine. OSUMC patients have completed the PROMIS-29 inventory, which includes information on cognitive functioning, overall functional status, and impact of cognitive symptoms on QoL.

SUMMARY:
Longitudinal study collecting retrospective and prospective data on treatments received and change in quality of life among patients with neurocognitive symptoms attending a Long COVID clinic

DETAILED DESCRIPTION:
Specific Aims:

1. Characterize pre-treatment quality of life and cognitive performance data for patients with Post-Acute Sequelae of COVID19 (PASC) and neurocognitive symptoms (PASC/NCS) seen at The Ohio State University Medical Center (OSUMC)
2. Describe treatment strategies deployed for these patients at the above institution.
3. Compare post-treatment quality of life and cognitive outcomes to pre-treatment values for these patients.

Significance and Impact:

Since the beginning of the epidemic, there have been 79 million COVID19 cases in the United States, and 480 million globally1. COVID19 survivors can suffer substantial long-term morbidity. Post-Acute Sequelae of COVID19 (PASC) is defined as persistent symptoms occurring weeks to months after infection with SARS-CoV-22. PASC is a multisystem disease with respiratory, cardiac, neurological, rheumatologic and other manifestations. In population-based studies, about 25% of patients report not having fully recovered 6-8 months after documented SARS-CoV-2 infection3. PASC is estimated to affect as many 17 million people worldwide4.

Neurocognitive symptoms in the setting of PASC (PASC/NCS) are seen 6 months after infection in 12-22% of COVID19 survivors5-8. They are associated with hypometabolism in brain areas controlling memory and executive function on brain imaging, and with atrophy in corresponding brain areas on post-mortem studies9-11. PASC/NCS has a significant impact on quality of life and functional ability, with 63% of affected patients reporting decreased quality of life12, and nearly half of previously employed patients unable to return to full-time work after 6 months13,14. Evidence suggests similar cellular mechanisms and patterns of neural injury between PASC/NCS and traumatic brain injury15-17.

Virtually all of the published literature to date on PASC/NCS is descriptive, focusing on epidemiology, phenotypes and putative mechanisms18-20. Given the high prevalence and impact of this condition, there is an urgent need for evidence-based strategies for managing and treating PASC/NCS. In our clinics, we have developed rehabilitative and pharmacologic strategies for treating such patients based on those used to aid recovery from brain injury. In this study, we will evaluate the impact of these strategies using standardized validated instruments to compare patient quality of life (QoL) and cognitive function (CF) on initial presentation and after treatment. This work will lay the groundwork for a larger study of an evidence-based treatment approach to PASC/NCS.

Research Strategy:

1. Institutional background

* OSUMC started a specialized multidisciplinary PASC clinic in March of 2021 to see patients suffering from persistent symptoms after COVID19 infection. The clinic is based in the Division of General Internal Medicine. To date we have seen 440 patients with PASC, of whom 177 had neurocognitive symptoms. Among the investigators, Dr. Grandominico is the PASC Clinic Director, and Drs. Friedberg and Schamess are the lead physicians.
* OSUMC patients have completed the PROMIS-29 inventory, which includes information on cognitive functioning, overall functional status, and impact of cognitive symptoms on QoL.

  1. Research plan
* Design: Study will include retrospective chart review and prospective data collection comparing pre- and post-treatment measures of symptom severity. OSU will include up to 440 patients for their retrospective chart review component and 100 patients for the prospective component.
* OSUMC will search its EMR for specified ICD-10 codes to identify patients with PASC/NCS seen in the past 12 months in the Post-COVID Recovery Clinic for potential inclusion in retrospective chart review and/or prospective study enrollment. For the prospective study data will be collected from patients until their 6-month post-treatment visit. The ICD-10 codes that associate with PASC/NCS have been identified in earlier work by our group.
* A designated research associate will review the charts from that institution to extract the following data for each subject:

  i. Pre-treatment QoL / cognitive function status using validated standard measures that are already collected for clinical purposes: PROMIS-29 scale, collected pre-treatment and 6 months post-treatment. Other data will include patient demographics, hospitalization (Y/N), ICU stay (Y/N), COVID19 vaccine history, comorbid conditions, and other signs and symptoms of PASC, comorbidities.

  i. Treatments recommended by clinician and initiated by patient, consisting of the following categories: cognitive rest, workplace accommodations, program of cognitive rehabilitation administered by a trained speech therapist, nutritional supplement (specify supplement), pharmacotherapy for PASC/NCS (specify medication). We will also record whether FMLA or other disability documentation was provided.

  i. Post-treatment QoL / cognitive function status using the same measures used for pre-treatment assessment.
* Data will be collected by authorized research staff from chart review and stored into Redcap, a secure data-sharing platform.
* Data will be analyzed by a biostatistician who will provide descriptive statistics and advise on handling of missing data.

  i. Extracted data will be analyzed for comparison of pre-treatment and post-treatment QoL / cognitive function status:
* Cumulative (for all subjects)
* By treatment category (see above)
* By treatment group: (a) supportive measures alone, (b) supportive measures plus cognitive rehabilitation, (c) supportive measures plus pharmacotherapy, and (d) combination of all three.
* This work will be submitted for publication at the Journal of the Neurological Sciences, Frontiers in Psychology, and the Journal of General Internal Medicine.

ELIGIBILITY:
Inclusion Criteria: For inclusion, patients had to have a diagnosis of Long COVID assigned by a PCRC provider and at least one of a prespecified set of ICD10 codes used by clinic providers to indicate neurologic symptoms. Since no diagnostic biomarkers or established criteria existed during the period of the study, Long COVID diagnosis was based on clinical judgement, taking into account the timing of symptom onset relative to acute COVID19 and the presence or absence of alternate diagnoses that might explain them.

-

Exclusion Criteria: Exclusion criteria were age under 18, failure to complete pre-visit PROMIS29 questionnaire, and absence of a Long COVID diagnosis or concurrent neurologic diagnosis.

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients recruited from the Post-COVID Recovery Clinic (PCRC) at the Ohio State University Wexner Medical Center (OSUWMC) between 10/12/2022 and 10/23/2023.
Sampling Method: Non-Probability Sample
Enrollment: 171 (Actual)
Dates: Start 2022-10-12 (Actual); Primary Completion 2024-03-31 (Actual); Study Completion 2024-04-01 (Actual)

PRIMARY OUTCOMES:
Change in quality of life using PROMIS26 questionnaire | 6 months
  The PROMIS29 is a well-validated measure of quality of life in multiple domains. Study subjects will complete PROMIS29 questionnaire at the first clinic visit, and again 6 months later. The outcome will consist of change in T-scores on the PROMIS29 from t=0 to t=6 months.
Change in PROMS20 T-scores | 6 months per patient
  Change in quality of life from pre-treatment to 6 months after initiating multimodality treatment in Post-CIVD Recovery Clinic. The PROMIS29 is a well-validated measure of quality of life in multiple domains.

CONTACTS AND LOCATIONS:
Locations (1):
- The Ohio State University Wexner Medical Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: Undecided
We need to better understand the aim of data sharing and how to go about it.